CLINICAL TRIAL: NCT06982196
Title: Multicenter, Randomized, Double-blinded，Controlled Clinical Study to Evaluate the Efficacy and Safety of Sulodexide in Controlling the Recurrence of Psoriasis
Brief Title: Sulodexide in Controlling the Recurrence of Psoriasis
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20242407-C-1
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-12

CONDITIONS: Psoriasis (PsO); Randomised Controlled Trial
Keywords: Randomized controlled trials
MeSH Terms: conditions — Psoriasis | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sulodexide Group (Experimental): Participants in this group will receive oral sulodexide soft capsules (manufactured by Alfa Wassermann, Italy; approval number H20140119, specification 250 LSU) after discontinuing secukinumab. The dosing regimen is 1 capsule twice daily for 120 consecutive days or until psoriasis relapse is confirmed. Sulodexide, a vascular protective agent, aims to prolong psoriasis recurrence by improving vascular endothelial barrier function. During the study, disease relapse (assessed via PASI scores) and safety indicators (e.g., adverse events, laboratory tests) will be regularly monitored.
  Interventions: Drug: Sulodexide
- Placebo Comparator Group (Placebo Comparator): Participants in this group will receive matching placebo capsules orally after discontinuing secukinumab. The dosing regimen is 1 capsule twice daily for 120 consecutive days or until psoriasis relapse is confirmed. The placebo capsules are identical in appearance and packaging to the active sulodexide capsules but contain no active pharmaceutical ingredients. This group serves as a control to evaluate the efficacy of sulodexide in delaying psoriasis recurrence. Disease relapse (assessed via PASIscores) and safety indicators (e.g., adverse events, laboratory tests) will be monitored at the same intervals as the experimental group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulodexide — Sulodexide group：Starting after the last injection of secukinumab, oral treatment with sulodexide soft capsule (Alpha Weissmann Pharmaceuticals, Italy, approval number H20140119, specification 250 LSU) was given as 1 tab bid for 120 days or discontinued after judged to be a relapse.
  Other Names: Vessel Due F (international brand)
  Arms: Sulodexide Group
Drug: Placebo — Control group: Oral treatment with placebo capsule, 1 tab bid starting after the last injection of secukinumab, discontinued after 120 days of continuous oral administration or judged to be discontinued for relapse.
  Other Names: Matching placebo for sulodexide soft capsules
  Arms: Placebo Comparator Group

SUMMARY:
This is a multicenter, randomized, double-blinded，controlled clinical trial. The purpose of the study is to evaluate the efficacy and safety of Sulodexide versus placebo in preventing psoriasis recurrence in patients with plaque psoriasis who have discontinued biologic therapy after achieving clinical cure.

DETAILED DESCRIPTION:
It was planned to include 160 patients with psoriasis vulgaris who met the inclusion criteria for discontinuation of biologics after reaching the standard of treatment and were randomised in a 1:1 ratio to receive oral treatment with sulodexide soft capsules or placebo capsules, respectively.

1. Sulodexide group： Starting after the last injection of secukinumab, oral treatment with sulodexide soft capsule (Alpha Weissmann Pharmaceuticals, Italy, approval number H20140119, specification 250 LSU) was given as 1 tab bid for 120 days or discontinued after judged to be a relapse;
2. Control group: Oral treatment with placebo capsule, 1 tab bid starting after the last injection of secukinumab, discontinued after 120 days of continuous oral administration or judged to be discontinued for relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18-65 years old and gender is not limited;
2. Clinical diagnosis consistent with moderate to severe plaque psoriasis;
3. After receiving standardised treatment with strychnicolizumab for 3 months to achieve complete clearing of skin lesions (in accordance with PASI 100 or PGA 0), and then continuing the treatment for 6 months without symptomatic relapse to satisfy the criteria for discontinuation of the drug and discontinuing strychnicolizumab (refer to the recommendations of 'Guidelines for the treatment of psoriasis with biologics in China (2021 edition)');
4. Voluntarily participate in the study and sign the informed consent form before the start of the study.

Exclusion Criteria:

1. Suffering from severe systemic or localised infections within the last 6 months;
2. Those with bleeding tendency or suffering from bleeding disorders;
3. The presence of malignant tumours, or postoperative tumour patients and those at high risk of tumours;
4. Have received or currently require treatment with other anticoagulant drugs such as sulodexide drugs within the last 9 months (e.g. argatroban, bivalirudin, dabigatran etexilate, desirudin, lepirudin, aspirin, etc.);
5. Treatment with other biological agents within the last 9 months;
6. Highly allergic or with a history of severe allergies; allergy to heparin or heparin analogues; or known/suspected allergy to one of the components of the investigational drug;
7. Infection with other diseases such as Human Immunodeficiency Virus (HIV);
8. Serious, progressive, uncontrolled disorders of vital organs and systems (including cardiovascular, hepatic, pulmonary, and renal) and other diseases that, in the opinion of the investigator, are not suitable for participation in the study in combination;
9. Clinically significant abnormal values on screening tests as determined by the investigator;
10. Pregnant women or women of childbearing potential who intend to become pregnant or breastfeeding during the trial period;
11. A positive serum or urine pregnancy test in a female of childbearing potential during the Screening Period;
12. Currently participating in another clinical study or have participated in another clinical study within 3 months;
13. Known presence of alcoholism, drug dependence, or psychiatric disorders
14. Known or suspected to be unable to complete the trial due to poor adherence;
15. Who, in the judgement of the investigator, are unsuitable for participation in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time of appearance of the first psoriatic skin lesion | 1 year
  This outcome measures the duration (in days) from the start of the study intervention (sulodexide or placebo) until the first identifiable recurrence of a characteristic psoriatic skin lesion in participants who had previously achieved complete clearance (PASI 100) with secukinumab therapy.

SECONDARY OUTCOMES:
Psoriasis lesion size and severity index score[PASI] | 1 year
  Psoriasis lesion size and severity index score
Dermatological Quality of Life Index[DLQI] | 1 year
  Dermatological Quality of Life Index
Self-Rating Anxiety Scale | 1 year
  The Self-Rating Anxiety Scale (SAS) is a validated 20-item questionnaire used to assess the severity of anxiety symptoms in participants. Each item is scored on a 4-point Likert scale (1 = "None or a little of the time" to 4 = "Most or all of the time"), with higher total scores indicating greater anxiety levels.
Self-Rating Depression Scale | 1 year
  The Self-Rating Depression Scale (SDS) is a widely used psychological assessment tool designed to measure the intensity and presence of depressive symptoms in individuals.
Adverse Events [AEs] | 1 year
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Principal Investigator — xjjing Hospital
Locations (1):
- xjjing Hospital, Xi'an, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffiths CEM, Armstrong AW, Gudjonsson JE, Barker JNWN. Psoriasis. Lancet. 2021 Apr 3;397(10281):1301-1315. doi: 10.1016/S0140-6736(20)32549-6. PMID 33812489
- [Background] Armstrong AW, Read C. Pathophysiology, Clinical Presentation, and Treatment of Psoriasis: A Review. JAMA. 2020 May 19;323(19):1945-1960. doi: 10.1001/jama.2020.4006. PMID 32427307
- [Background] Tian D, Lai Y. The Relapse of Psoriasis: Mechanisms and Mysteries. JID Innov. 2022 Mar 9;2(3):100116. doi: 10.1016/j.xjidi.2022.100116. eCollection 2022 May. PMID 35601055
- [Background] Chen L, Shen Z. Tissue-resident memory T cells and their biological characteristics in the recurrence of inflammatory skin disorders. Cell Mol Immunol. 2020 Jan;17(1):64-75. doi: 10.1038/s41423-019-0291-4. Epub 2019 Oct 8. PMID 31595056
- [Background] Yelamos O, Alejo B, Ertekin SS, Villa-Crespo L, Zamora-Barquero S, Martinez N, Dominguez M, Iglesias P, Herrero A, Malvehy J, Puig S. Non-invasive clinical and microscopic evaluation of the response to treatment with clobetasol cream vs. calcipotriol/betamethasone dipropionate foam in mild to moderate plaque psoriasis: an investigator-initiated, phase IV, unicentric, open, randomized clinical trial. J Eur Acad Dermatol Venereol. 2021 Jan;35(1):143-149. doi: 10.1111/jdv.16559. Epub 2020 Jul 6. PMID 32365242
- [Background] Zhu Z, Chen J, Lin Y, Zhang C, Li W, Qiao H, Fu M, Dang E, Wang G. Aryl Hydrocarbon Receptor in Cutaneous Vascular Endothelial Cells Restricts Psoriasis Development by Negatively Regulating Neutrophil Recruitment. J Invest Dermatol. 2020 Jun;140(6):1233-1243.e9. doi: 10.1016/j.jid.2019.11.022. Epub 2019 Dec 30. PMID 31899186
- [Background] Chen J, Zhu Z, Li Q, Lin Y, Dang E, Meng H, Sha N, Bai H, Wang G, An S, Shao S. Neutrophils Enhance Cutaneous Vascular Dilation and Permeability to Aggravate Psoriasis by Releasing Matrix Metallopeptidase 9. J Invest Dermatol. 2021 Apr;141(4):787-799. doi: 10.1016/j.jid.2020.07.028. Epub 2020 Sep 2. PMID 32888954
- [Background] Li Q, Zhu Z, Wang L, Lin Y, Fang H, Lei J, Cao T, Wang G, Dang E. Single-cell transcriptome profiling reveals vascular endothelial cell heterogeneity in human skin. Theranostics. 2021 Apr 19;11(13):6461-6476. doi: 10.7150/thno.54917. eCollection 2021. PMID 33995668
- [Background] Li Q, Shao S, Zhu Z, Chen J, Hao J, Bai Y, Li B, Dang E, Wang G. An IGFBP7hi endothelial cell subset drives T cell extravasation in psoriasis via endothelial glycocalyx degradation. J Clin Invest. 2023 May 1;133(9):e160451. doi: 10.1172/JCI160451. PMID 36917196
- See also: PubMed is a free search engine maintained by the U.S. National Library of Medicine (NLM). It provides access to over 38 million citations from MEDLINE, life science journals, and online books, often linking to full - text articles on PubMed Central or pu — https://pubmed.ncbi.nlm.nih.gov/